CLINICAL TRIAL: NCT00832637
Title: Gemcitabine and Cisplatin With Erlotinib in Hepatocellular Carcinoma (HCC) and Biliary Tree Cancer (BTC) (Intra- and Extra-hepatic Cholangiocarcinoma, Bile Duct Cancer, Adenocarcinoma of the Ampulla of Vater and Gallbladder Carcinoma)
Brief Title: Gemcitabine, Oxaliplatin, Tarceva &/or Cisplatin in HCC & Biliary Tree Cancers
Acronym: Gem-ox
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST OX-05-024; NCI-2011-02729 (Registry Identifier: NCI Clinical Trial Reporting Program); B9E-US-X467 (Other Grant/Funding Number: Eli Lilly)
Record Dates: First submitted 2009-01-13; First posted 2009-01-30 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Hepatocellular Carcinoma; Cholangiocellular Carcinoma; Cholangiocarcinoma of the Extrahepatic Bile Duct; Bile Duct Cancer; Periampullary Adenocarcinoma; Gallbladder Cancer; Extrahepatic Bile Duct Cancer
Keywords: Liver; Gallbladder; Bile duct; Gemzar; Eloxatin; Tarceva; erlotinib; Gem-ox
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Cisplatin; Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Cisplatin, Erlotinib (Experimental): A combination of Cisplatin at 40 mg/m2 + Gemcitabine at 1000 mg/m2, every 28 days + Erlotinib 100 mg daily, orally. Cycles will be repeated every four weeks.
  Interventions: Drug: Cisplatin; Drug: Erlotinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Cisplatin — Cisplatin is administered intravenously at 40 mg/m2 on day 1 and day 15, every 28 days. Cisplatin is administered following Gemcitabine. Cisplatin administration should occur with hydration with normal saline at 250 mL/ hour for at least 4 hours before and during Cisplatin administration. Additionally, Cisplatin administration should be preceded by osmotic diuresis with Mannitol 25%, 12.5 grams.
  Other Names: Platinol®
Drug: Erlotinib — 100 mg orally daily. For grade 3 or 4 skin rash, erlotinib should be held until resolution of the rash to no more than grade 1 before resumption of erlotinib.
  Other Names: Tarceva®
Drug: Gemcitabine — Gemcitabine is administered intravenously at 1000 mg/m2 on day 1 and 15, every 28 days. The clinical formulation is supplied in a sterile form for intravenous use only. Vials of gemcitabine contain either 200 mg or 1 g of gemcitabine hydrochloride (HCl )(expressed as free base) formulated with mannitol (200 mg or 1 g, respectively) and sodium acetate (12.5 mg or 62.5 mg, respectively) as a sterile lyophilized powder. Hydrochloric acid and/or sodium hydroxide may have been added for pH adjustment.
  Other Names: Gemzar®

SUMMARY:
This is a single arm phase II trial of Gemcitabine and Oxaliplatin (Gem-Ox) with Erlotinib (Tarceva) for the treatment of hepatocellular carcinoma (HCC) and biliary tree cancer (BTC) patients with platelet counts 100,000/µL. The purpose of this study is to determine the tumor control rate following treatment with GEM-OX combined with Tarceva in patients with HCC. Tumor control rate is defined as the percentage of patients achieving a complete response, partial response, or stable disease at 24 weeks following treatment.

DETAILED DESCRIPTION:
The incidence and mortality of HCC has increased in the United States. Promising responses have been observed in HCC patients treated with gemcitabine and cisplatin, inclusing good disease stabilization and progression free survival. Cisplatin-gemcitabine enhances the cytotoxicity of cisplatin by increasing the formation of cytotoxic platinum DNA adducts. Similarly, Oxaliplatin also has DNA cross linkage properties and one could assume that its combination with gemcitabine is likely to potentiate the cytotoxicity of the latter. Erlotinib has also been reported to result in clinical benefit in HCC and BTC patients. Based on these prior findings, we embarked on this phase II protocol of gemcitabine, oxaliplatin, and erlotinib in HCC and BTC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC) or biliary tree cancer (BTC:: intra- and extra-hepatic cholanciocarcinoma, bile duct cancer, adenocarcinoma of the Ampulla of Vater and/or gallbladder carcinoma).
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST).
* Age 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2
* Adequate bone marrow as evidenced by:

  * Absolute neutrophil count (ANC) > 1,500/L.
  * Platelet count > 100,000/L.
  * Absence of a regular red blood cell transfusion requirement.
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL.
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin 1.5x Upper Limit of Normal (ULN).
  * Alkaline phosphatase < 3x ULN for the reference lab (< 5x ULN for patients with known hepatic metastases).
  * Serum glutamic-oxaloacetic transaminase (SGOT)/ serum glutamic-pyruvic transaminase (SGPT) < 3x ULN for the reference lab (< 5x ULN for patients with known hepatic metastases).
* Patients must have a life expectancy of 12 weeks.
* Patients must be recovered from both acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy.
* Patients of childbearing potential agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method).

Exclusion Criteria:

A patient may not be enrolled in the trial if any of the following criteria are met:

* Patients with an active infection or with a fever > 38.50 degrees Celcius within 3 days of the first scheduled day of protocol treatment.
* Patients with active central nervous system (CNS) metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for 3 weeks are eligible for the trial.
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current prostate serum antigen (PSA) of < 1.0 mg/dL on 2 successive evaluations at least 3 months apart, with the most recent evaluation within 4 weeks of entry.
* Patients with prior treatment or known hypersensitivity to any of the components of oxaliplatin or gemcitabine.
* Patients who have received chemotherapy within 30 days of the first scheduled day of protocol treatment.
* Patients who received radiotherapy to more than 25% of their bone marrow; or patients who received any radiotherapy within 4 weeks of entry.
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).
* Peripheral neuropathy Grade 2.
* Patients who are pregnant or lactating.
* Patients with a life expectancy of less than 12 weeks.
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator, likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* Patients with any of the following laboratory parameters:

  * Abnormal hematological values with ANC < 1500/mm3, thrombocytopenia < 99,000.
  * Impaired renal function with a serum creatinine > 1.5x ULN.
  * Serum bilirubin > 1.5xULN.
  * Albumin < 2.5 mg/dl.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.
* History of allogeneic transplant.
* Known human immunodeficiency virus (HIV).
* Clinically significant heart disease defined as New York Heart Association (NYHA) class 3 or 4 heart disease.
* Known or existing uncontrolled coagulopathy.
* Patients with severe medical problems such as uncontrolled diabetes or chronically debilitating diseases that the investigator feels might compromise the study participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Patt, MD, Principal Investigator — University of New Mexico; Ari D Baron, MD, Principal Investigator — California Pacific Medical Center
Locations (2):
- United States (2):
  - California Pacific Medical Center, San Francisco, California
  - University of New Mexico Cancer Center, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine, Cisplatin, Erlotinib: Cisplatin at a dose of 40 mg/m2 q 2 weeks along with gemcitabine, 1000mg/m2, and erlotinib 100 mg daily PO.
  Cisplatin: Cisplatin 40 mg/ m2 on day 1 and day 15 in patients treated with Gem + Cis, with Cisplatin to be given following Gemcitabine. Cisplatin administration should be given along with hydration with NS at 250 mL/ hour for at least 4 hours pre-and during Cisplatin administration. Additionally, Cisplatin administration should be preceded by osmotic diuresis with Mannitol 25%, 12.5 grams.
  Erlotinib: 100 mg orally daily.
  Gemcitabine: 1000 mg/m2 on Days 1, 15 every 28 days. The clinical formulation is supplied in a sterile form for intravenous use only. Vials of gemcitabine contain either 200 mg or 1 g of gemcitabine HCl (expressed as free base) formulated with mannitol (200 mg or 1 g, respectively) and sodium acetate (12.5 mg or 62.5 mg, respectively) as a sterile lyophilized powder. Hydrochloric acid and/or sodium hydroxide may have been added for pH adjustment.
Period: Overall Study
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 59 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Tumor Control Rate
Description: Rate of tumor control is defined as the percentage of patients achieving a complete response (CR) + partial response (PR) + stable disease (SD) at 24 weeks following treatment.
  Response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 24 weeks
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Number analyzed (Participants) | 33
percentage of evaluable participants
  Complete response (CR) | 0
  Partial response (PR) | 7.1
  Stable disease (SD) | 53.6
  CR + PR + SD | 60.7

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of patients achieving a complete response (CR) + partial response (PR) at 24 weeks following treatment.
  Response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 24 weeks
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Number analyzed (Participants) | 28
percentage of evaluable participants
  Complete response (CR) | 0
  Partial response (PR) | 7.1
  CR + PR | 7.1

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: The time from treatment initiation to disease progression. Progression is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI): Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Number analyzed (Participants) | 33
weeks | 22 [18 to 78]

4. Secondary Outcome: Median Survival Time (MST)
Description: Survival is defined as the time from treatment initiation to death by any cause
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Number analyzed (Participants) | 33
weeks | 28 [21 to 53]

5. Secondary Outcome: Toxicity
Description: Toxicity will be evaluated per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Frequency and severity of adverse events will be tabulated using counts of frequently occurring, serious and severe events of interest (i.e. Grade 3 and Grade 4 adverse events).
Time Frame: Patients are followed for at least one month following end of on-study treatment. All patients who discontinue the trial secondary to an adverse event are followed until resolution, stabilization or return to a baseline condition. An average of 24 weeks
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Number analyzed (Participants) | 33
participants
  Anemia | 2
  Neutropenia | 7
  Neutropenic Fever | 2
  Thrombocytopenia | 6
  Diarrhea | 4
  Abdominal Pain | 2
  Renal Failure | 1
  Dermatitis (acneiform) | 3
  Peripheral neuropathy | 1
  Metabolic syndrome | 2
  Cerebral hemorrhage | 1

ADVERSE EVENTS:
Time Frame: Patients are followed for at least one month following end of on-study treatment. All patients who discontinue the trial secondary to an adverse event are followed until resolution, stabilization or return to a baseline condition, an average of 24 weeks.
Arm/Group | Gemcitabine, Cisplatin, Erlotinib
Serious Adverse Events (participants affected / at risk) | 17/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Cisplatin, Erlotinib (N=33)
Hypersensitivity reaction (Immune system disorders) | 1 (1)
Hemolysis (Red blood cell destruction) (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (3)
Anorexia (Loss of appetite) (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastritis (Stomach lining inflammation) (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Hypokalemia (Low potassium level in blood) (Investigations) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Abdominal pain (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Death (General disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Cisplatin, Erlotinib (N=33)
Rhinitis (Runny nose) (General disorders) | 5 (12)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (12)
Hemolysis (Red blood cell destruction) (Blood and lymphatic system disorders) | 7 (7)
Leukocytes decreased (Blood and lymphatic system disorders) | 7 (10)
Neutrophils decreased (Blood and lymphatic system disorders) | 7 (18)
Platelet count decreased (Blood and lymphatic system disorders) | 14 (44)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 22 (27)
Fever (General disorders) | 8 (9)
Weight Loss (General disorders) | 5 (6)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 2 (3)
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Acne (Skin and subcutaneous tissue disorders) | 9 (12)
Desquamating rash (Skin and subcutaneous tissue disorders) | 9 (9)
Abdominal distention (Gastrointestinal disorders) | 3 (3)
Anorexia (Loss of appetite) (Gastrointestinal disorders) | 10 (10)
Ascites (Accumulation of fluid in the abdomen) (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (9)
Dehydration (Gastrointestinal disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 18 (22)
Gastritis (Stomach lining inflammation) (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (19)
Vomiting (Gastrointestinal disorders) | 11 (14)
Epistaxis (Nosebleed) (General disorders) | 3 (3)
Febrile neutropenia (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Edema: limbs (General disorders) | 3 (5)
Edema: trunk/genital (General disorders) | 2 (3)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Hyperbilirubinemia (High level of bilirubin) (Investigations) | 6 (10)
Hyperglycemia (High glucose level in blood) (Investigations) | 3 (4)
Hypoalbuminemia (Low level of albumin in blood) (Investigations) | 4 (8)
Hypocalcemia (Low calcium level in blood) (Investigations) | 3 (5)
ypocalcemia (Low calcium level in blood) (Investigations) | 3 (5)
Hypokalemia (Low potassium level in blood) (Investigations) | 5 (9)
Hypomagnesemia (Low magnesium level in blood) (Investigations) | 3 (4)
Hyponatremia (Low sodium level in blood) (Investigations) | 4 (5)
Anxiety (Nervous system disorders) | 3 (3)
Confusion (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (4)
Insomnia (Nervous system disorders) | 7 (7)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5)
Abdominal pain (General disorders) | 5 (8)
Extremity - Limb pain (General disorders) | 2 (2)
Neck Pain (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes